CLINICAL TRIAL: NCT05529797
Title: Effect of a Single Virtual Reality Exposure on Depressive Symptoms (Veovita-VR): Randomized Controlled Trial
Brief Title: Effect of a Single Virtual Reality Exposure on Depressive Symptoms (Veovita-VR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Veovita-VR
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Depression
Keywords: Virtual Reality; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Veovita-VR (Experimental): Participants receive one VR session with positive emotional stimuli and positive behavioral activation.
  Interventions: Other: Veovita-VR
- Care as Usual (No Intervention): Participants receive CAU.

INTERVENTIONS:
Other: Veovita-VR — Veovita-VR is a VR intervention with positive emotional stimuli and positive behavioral activation designed to reduce depressive symptoms in people with at least moderate depressive symptoms. In the VR session, the participants stay in a beautiful environment (island, sandy beach, beautiful scenery). They can engage in activities that are perceived as positive (climbing, treasure hunting, listening to music, building sandcastles). The session has a length of approx. 30 minutes. Participants are free to continue to engage with any treatment they require during the duration of the study.
  Arms: Veovita-VR

SUMMARY:
The trial aims to evaluate the effectiveness of a novel virtual reality (VR) intervention (Veovita-VR) designed to expose people with at least moderate depressive symptoms to positive emotional stimuli and positive behavioral activation, thereby reducing depressive symptoms. Therefore, 128 adults with at least moderate depressive symptoms (operationalized as a Patient Health Questionnaire (PHQ-9) score ≥ 10) will be recruited and randomized into two groups: (1) a control group that may undergo depression treatment (Care-as-Usual, CAU) and receive access to Veovita-VR 5 weeks post-baseline (i.e., CAU control group), or (2) to an intervention group that receives one Veovita-VR session immediately after randomization and may also use CAU. The primary endpoint is depressive symptom level as assessed with the Patient Health Questionnaire (PHQ-9) 4 weeks post-baseline. Additionally, depressive symptoms (PHQ-9) will be assessed 1 week post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* PHQ-9 score ≥ 10

Exclusion Criteria:

* apparent mental health problems other than depression (e.g., diagnosis of substance use disorder, psychotic disorder or bipolar disorder)
* acute suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 4 weeks after baseline
  The PHQ-9 is a well-validated nine-item self-report questionnaire developed to score each of the nine DSM-IV criteria for major depressive disorder on a 4-point Likert scale, from "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 1 week after baseline
  The PHQ-9 is a well-validated nine-item self-report questionnaire developed to score each of the nine DSM-IV criteria for major depressive disorder on a 4-point Likert scale, from "0" (not at all) to "3" (nearly every day).

CONTACTS AND LOCATIONS:
Overall Officials: Gitta Jacob, PD Dr., Principal Investigator — Gaia AG
Locations (1):
- Gaia AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No